CLINICAL TRIAL: NCT01162213
Title: Effects of Lychee Fruit Extract on Vascular Function and Inflammation in Postmenopausal Women: a Double-Blind, Crossover Study
Brief Title: Pilot Study of Lychee Fruit Extract to Promote Cardiovascular Health
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Robert M Hackman, Nutrition Department, University of California, Davis
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 200916915-2
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Cardiovascular Health
Keywords: Postmenopausal Women; Healthy Males; Cardiovascular; Flavanols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 100 mg of Lychee fruit extract (Experimental)
  Interventions: Dietary Supplement: Lychee Fruit Extract
- 200 mg of Lychee fruit extract (Experimental)
  Interventions: Dietary Supplement: Lychee Fruit Extract
- 600 mg of Lychee fruit extract (Experimental)
  Interventions: Dietary Supplement: Lychee Fruit Extract
- 2000 mg of Lychee fruit extract (Experimental)
  Interventions: Dietary Supplement: Lychee Fruit Extract

INTERVENTIONS:
Dietary Supplement: Lychee Fruit Extract — placebo or 100, 200 and 600 mg of lychee fruit extract for 2 weeks with one week washout period between treatments 2000 mg of lychee fruit extract given at a single visit

SUMMARY:
The investigators hypothesize that acute and short term consumption of a lychee fruit extract, particularly rich in low molecular weight dietary flavanols, will improve vascular function and reduce platelet reactivity.

DETAILED DESCRIPTION:
Several large-scale epidemiologic studies have indicated that chronic consumption of flavonoid-rich foods appear to be associated with decreased risk for several chronic diseases including cancer, diabetes, cardiovascular disease, and stroke. In humans, consumption of several flavonoid-rich foods and beverages, such as berries, teas, cocoa, and grapes have been reported to improve vascular endothelial function and decrease platelet reactivity. Previous work at UC Davis by Dr. Keen and colleagues has helped define the role of flavanols in vascular function, and has used a flavanol-rich cocoa extract as the test material. In this proposed study, we seek to explore the role of a lychee fruit extract rich in flavanols, and its effects of vascular and metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Female Age 52 to 65 yrs.
* Male Age 18 to 35 yrs.
* Female and male >110 pounds
* Lack of menses in the last year and FSH 23-116.3 mIU/mL
* Subject is willing and able to comply with the study protocols.
* Subject is willing to consume the lychee fruit extract or placebo capsule twice a day.
* BMI 20-35 kg/m2

Exclusion Criteria:

* Physical signs of health impairment
* Weight < 110 pounds
* BMI >35 kg/m2
* Blood Pressure > 140/90 mm Hg
* Diabetes
* Inability to properly place or wear the PAT probes or abnormal measurements on pre-screening PAT
* Abnormal clinical laboratory test (CBC, comprehensive metabolic panel, etc.) if determined to be clinically significant by Dr. M. Eric Gershwin.
* PFA-100 readings 10% outside of normal reference range (normal reference range for ADP-Collagen cartridge: 71-118 sec; Epinephrine-Collagen cartridge: 94-193 sec).
* Inflammatory disorders (e.g. rheumatoid arthritis)
* Malabsorption
* Treatment with corticosteroids, hypolipidemic and anti-inflammatory drugs
* Renal or liver disease
* History of cancer
* Heart disease, which includes cardiovascular events and Stroke
* Cushing's syndrome
* History of psychiatric disorders i.e. schizophrenia or bi-polar or depression treated with antidepressants within the last 1 year.
* Anxiety medications
* Routine use of prescription drugs or over-the counter medications, which may potentially modulate the outcome of this study; including antibiotics, aspirin and aspirin-containing formulations, COX-2 inhibitors, antihistamines, corticosteroids
* Asthma (can be worsened by mild to moderate food allergies)
* Indications of substance or alcohol abuse within the last 3 years
* Multi-vitamin and mineral use other than a general formula, once per day tablet
* Use of herbal or plant-based supplements; omega-3 fatty acids, and fish oils in the past 3-6 months, and unwilling to discontinue use while participating in the study
* Alcohol consumption > 1 oz/day (2 beers/day or 2 glasses of wine/ day, 1 drink of hard liquor/day)
* Allergies to fruit
* Chronic/routine high-intensity exercise
* Smoking or actively in smoking cessation therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Peripheral Arterial Tonometry | 0, 2 and 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Hackman, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Ragle Human Nutrition Research Center, Davis, California, United States